CLINICAL TRIAL: NCT07061015
Title: Evaluation Of Different Motor Driven Osseodensification Techniques Used For Implant Placement In Posteriorly Atrophied Mandible Of Osteoporotic Patients
Brief Title: Efficacy of Different Osseodensification Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A01030123
Record Dates: First submitted 2025-06-22; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Osseodensification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- osseodensifying burs (Active Comparator): osseodensifying burs are used in reverse motion .
  Interventions: Procedure: osseodenification with osseodensifying burs
- reverse drilling (Active Comparator): using conventional implant drills in reverse motion(anti clock wise)
  Interventions: Procedure: reverse drilling
- rotary expanders (Active Comparator): using rotary expanders in clock wise motion
  Interventions: Procedure: rotary expanders

INTERVENTIONS:
Procedure: osseodenification with osseodensifying burs — different osseodensification techniques to be studied
  Arms: osseodensifying burs
Procedure: reverse drilling — using the conventional drills in reverse mode
  Arms: reverse drilling
Procedure: rotary expanders — expanders in clockwise direction
  Arms: rotary expanders

SUMMARY:
different possible osseodensification techniques used to improve bone density around dental implants, using either ] osseodensifying drills, reverse drilling of conventional drills, and rotary expanders.

DETAILED DESCRIPTION:
the study include 3 groups with different implant drilling protocols; group 1 where osseodensifying burs are used, group 2 where conventional drills with reverse motion are used, group 3 where rotary expanders are used

ELIGIBILITY:
Inclusion Criteria:

* · Adult osteoporotic female patients confirmed by CBCT grey values ranging from 290 to 420 HU, with age range 45-60 years.

  * Patients should be free from any other systemic diseases, according to ASA classifications (American society of Anesthesiologists).
  * Patients of single or multiple missing teeth in the posterior mandible.
  * A ridge width of 4mm and a height of > 8mm above the roof of Inferior Alveolar canal.
  * No buccal concavities were present at the planned implant site

Exclusion Criteria:

* · Poor oral hygiene.

  * Heavy smoker (more than 20 cigarettes /day),or alcoholic abusing patients.
  * Radiation therapy to the head and neck region, or chemotherapy in the last 6 months prior to the implant placement.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
peri implant bone density | 12 months
  through ROI (region of interest) to measure Grey scale on Cone beam computed tomography CBCT
implant stability quotient | 12 months
  ISQ (implant stability quotient) using osstell device
alveolar ridge dimension changes | 12 months
  with cone beam computed tomography CBCT in coronal and sagittal cuts, in millimeters mm .

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed MZ M Zaghlol Amer, Professor, Study Director — Mansoura University
Locations (1):
- Delta university for science and technology, Al Mansurah, Daqhlia, Egypt